CLINICAL TRIAL: NCT01819129
Title: Efficacy and Safety of FIAsp Compared to Insulin Aspart in Combination With Insulin Glargine and Metformin in Adults With Type 2 Diabetes
Acronym: onset® 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-3853; 2010-024051-93 (EudraCT Number); U1111-1118-2509 (Other: WHO); CTRI/2014/01/004285 (Registry Identifier: Clinical Trials Registry - India (CTRI))
Record Dates: First submitted 2013-03-21; First posted 2013-03-27 (Estimated); Results first posted 2017-12-05 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Faster-acting insulin aspart (FIAsp) (Experimental): Meal time faster-acting insulin aspart is given in combination with once daily insulin glargine and metformin in a basal-bolus regimen. Insulin glargine and metformin treatment are open labelled background medication.
  Interventions: Drug: Faster-acting insulin aspart; Drug: Insulin glargine
- Insulin aspart (Active Comparator): Meal time insulin aspart is given in combination with once daily insulin glargine and metformin in a basal-bolus regimen. Insulin glargine and metformin treatment are open labelled background medication.
  Interventions: Drug: Insulin aspart; Drug: Insulin glargine

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Mealtime FIAsp administered subcutaneously (s.c., under the skin). Dose individually adjusted.
  Arms: Faster-acting insulin aspart (FIAsp)
Drug: Insulin aspart — Mealtime insulin aspart administered subcutaneously (s.c., under the skin). Dose individually adjusted.
  Arms: Insulin aspart
Drug: Insulin glargine — Administered s.c. once daily at subjects' pre-trial dose. Subjects will continue their metformin treatment without changing the frequency or dose throughout the trial.

SUMMARY:
This trial is conducted in Asia, Europe and North America. The aim of the trial is to compare FIAsp (faster-acting insulin aspart) to insulin aspart, both in combination with insulin glargine and metformin in adults with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria: - Type 2 diabetes (diagnosed clinically) for 6 months or longer at time of screening (visit 1) - Treated with basal insulin for at least 6 months prior to screening (visit 1) - Current once daily treatment with insulin NPH (Neutral Protamine Hagedorn), insulin detemir or glargine for at least 3 months prior to the screening visit (visit 1) - Current treatment with: a. metformin with unchanged dosing for at least 3 months prior to screening (visit 1). The metformin dose must be at least 1000 mg or b. metformin in combination with sulfonylurea (SU) or glinide or DPP-IV (dipeptidyl peptidase-4) inhibitors and/or alpha-glucosidase inhibitors (AGI) with unchanged dosing for at least 3 months prior to screening (visit 1). The metformin dose must be at least 1000 mg - HbA1c by central laboratory: a. 7.0 - 9.5% (53 - 80 mmol/mol) (both inclusive) in the metformin group at the screening visit (visit 1) or b. 7.0 - 9.0% (53 - 75 mmol/mol) (both inclusive) in the metformin + other OAD (oral antidiabetic drug) (SU, glinide, DDP-IV inhibitors, AGI) combination group at the screening visit (visit 1) - Body mass index (BMI) equal to or below 40.0 kg/m^2 Exclusion Criteria: - Any use of bolus insulin, except short-term use due to intermittent illness (no longer than 14 days consecutive treatment) and not 3 months prior to the screening visit (visit 1) - Use of GLP-1 (glucagon-like peptide-1) agonists and/or TZDs within the last 3 months prior to screening (visit 1) - Recurrent severe hypoglycaemia (more than 1 severe hypoglycaemic event during the last 12 months) or hypoglycaemic unawareness as judged by the Investigator or hospitalisation for diabetic ketoacidosis during the previous 6 months prior to screening (visit 1) - Cardiovascular disease, within the last 6 months prior to screening (visit 1), defined as: stroke, decompensated heart failure New York Heart Association (NYHA) class III or IV, myocardial infarction, unstable angina pectoris or coronary arterial bypass graft or angioplasty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 881 (Actual)
Dates: Start 2013-09-09 (Actual); Primary Completion 2015-01-22 (Actual); Study Completion 2015-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (125):
- United States (71):
  - Novo Nordisk Investigational Site, Glendale, Arizona
  - Novo Nordisk Investigational Site, Mesa, Arizona
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Tempe, Arizona
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Greenbrae, California
  - Novo Nordisk Investigational Site, Lomita, California
  - Novo Nordisk Investigational Site, Northridge, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, San Ramon, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Boynton Beach, Florida
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Cooper City, Florida
  - Novo Nordisk Investigational Site, Fort Lauderdale, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Decatur, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Avon, Illinois
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Muncie, Indiana
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Madisonville, Kentucky
  - Novo Nordisk Investigational Site, Paducah, Kentucky
  - Novo Nordisk Investigational Site, Monroe, Louisiana
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Detroit, Michigan
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, Jefferson City, Missouri
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, Butte, Montana
  - Novo Nordisk Investigational Site, Elkhorn, Nebraska
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Mineola, New York
  - Novo Nordisk Investigational Site, New Windsor, New York
  - Novo Nordisk Investigational Site, North Massapequa, New York
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, Hickory, North Carolina
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Carlisle, Ohio
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Dayton, Ohio
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Mason, Ohio
  - Novo Nordisk Investigational Site, East Providence, Rhode Island
  - Novo Nordisk Investigational Site, Gaffney, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Spring Hill, Tennessee
  - Novo Nordisk Investigational Site, Tullahoma, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Hurst, Texas
  - Novo Nordisk Investigational Site, Plano, Texas
  - Novo Nordisk Investigational Site, Murray, Utah
  - Novo Nordisk Investigational Site, Midlothian, Virginia
  - Novo Nordisk Investigational Site, Port Orchard, Washington
  - Novo Nordisk Investigational Site, Kenosha, Wisconsin
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Canada (11):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Surrey, British Columbia
  - Novo Nordisk Investigational Site, Mount Pearl, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, St. John's, Newfoundland and Labrador
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Thunder Bay, Ontario
  - Novo Nordisk Investigational Site, Waterloo, Ontario
  - Novo Nordisk Investigational Site, Mirabel, Quebec
  - Novo Nordisk Investigational Site, Montreal, Quebec
  - Novo Nordisk Investigational Site, Saint Romuald, Quebec
  - Novo Nordisk Investigational Site, Québec
- Croatia (7):
  - Novo Nordisk Investigational Site, Čakovec
  - Novo Nordisk Investigational Site, Karlovac
  - Novo Nordisk Investigational Site, Osijek
  - Novo Nordisk Investigational Site, Slavonski Brod
  - Novo Nordisk Investigational Site, Split
  - Novo Nordisk Investigational Site, Varaždin
  - Novo Nordisk Investigational Site, Zagreb
- India (7):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Delhi, New Delhi
  - Novo Nordisk Investigational Site, Bhubaneswar, Odisha
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
- Israel (6):
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Kfar Saba
  - Novo Nordisk Investigational Site, Rehovot
  - Novo Nordisk Investigational Site, Rishon LeZiyyon
- Novo Nordisk Investigational Site, Ponce, Puerto Rico
- Russia (6):
  - Novo Nordisk Investigational Site, Kursk
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saint-Petesburg
  - Novo Nordisk Investigational Site, Stavropol
- Serbia (3):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Niš
  - Novo Nordisk Investigational Site, Zaječar
- Slovakia (4):
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Lučenec
  - Novo Nordisk Investigational Site, Trnava
  - Novo Nordisk Investigational Site, Žilina
- United Kingdom (9):
  - Novo Nordisk Investigational Site, Epworth
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Northampton
  - Novo Nordisk Investigational Site, Northwood
  - Novo Nordisk Investigational Site, Norwich
  - Novo Nordisk Investigational Site, Nuneaton
  - Novo Nordisk Investigational Site, Sidcup
  - Novo Nordisk Investigational Site, Stoke-on-Trent
  - Novo Nordisk Investigational Site, Wrexham

REFERENCES:
- [Result] Bowering K, Case C, Harvey J, Reeves M, Sampson M, Strzinek R, Bretler DM, Bang RB, Bode BW. Faster Aspart Versus Insulin Aspart as Part of a Basal-Bolus Regimen in Inadequately Controlled Type 2 Diabetes: The onset 2 Trial. Diabetes Care. 2017 Jul;40(7):951-957. doi: 10.2337/dc16-1770. Epub 2017 May 8. PMID 28483786
- [Result] Bode BW, Bowering K, Russell-Jones D. Response to Comment on Russell-Jones et al. Diabetes Care 2017;40:943-950. Comment on Bowering et al. Diabetes Care 2017;40:951-957. Diabetes Care. 2018 Mar;41(3):e29-e30. doi: 10.2337/dci17-0051. No abstract available. PMID 29463670
- [Result] Bowering K, Rodbard HW, Russell-Jones D, Bode B, Harris S, Piletic M, Heller S, Woo V, Babu V, Dethlefsen C, Mathieu C. Investigating the Association Between Baseline Characteristics (HbA1c and Body Mass Index) and Clinical Outcomes of Fast-Acting Insulin Aspart in People with Diabetes: A Post Hoc Analysis. Diabetes Ther. 2019 Feb;10(1):177-188. doi: 10.1007/s13300-018-0553-7. Epub 2018 Dec 13. PMID 30547388
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 150 sites, which were selected for recruitment, 128 sites in 9 countries enrolled subjects in the run-in period, of which 123 sites later assigned subjects to randomized treatment: Canada:9 sites; Croatia:6 sites; India:6 sites; Israel:6 sites; Russia:12 sites; Serbia:9 sites; Slovakia:5 sites; United Kingdom:7 sites; United States:63 sites.
Pre-assignment Details: The trial included an 8-week run-in period and a 26-week treatment period. During the run-in period, the subjects received insulin glargine along with metformin. In total, 881 subjects entered the run-in period, of these 192 subjects were run-in failures. Hence, 689 subjects entered the 26-week treatment period.
Groups:
- Faster Aspart: At randomization, all subjects started on 4 units of mealtime faster aspart (bolus insulin) in combination with once-daily subcutaneous (sc) injection of insulin glargine (basal insulin) and metformin (oral) in a basal-bolus regiment. Faster aspart was administered (sc) 0-2 minutes before each main meal and dose was titrated to the pre-prandial glycaemic target of 4.0-6.0 mmol/L (71-108 mg/dL) in a treat-to-target fashion according to the titration guideline. Dose adjustments were considered daily based on the pre-prandial and bedtime self-measured plasma glucose (SMPG) on the previous day. The dose adjustments were -1 or +1 if the pre-prandial or bedtime plasma glucose was <4.0 mmol/L or >6.0 mmol/L respectively. Basal insulin dose adjustments were allowed when needed. Metformin treatment continued without changing the frequency or dose.
- NovoRapid: At randomization, all subjects started on 4 units of mealtime NovoRapid®/NovoLog® (insulin aspart; bolus insulin) in combination with once-daily sc injection of insulin glargine (basal insulin) and metformin (oral) in a basal-bolus regimen. NovoRapid®/ NovoLog® was administered (sc) 0-2 minutes before each main meal, was titrated to the pre-prandial glycaemic target of 4.0-6.0 mmol/L (71-108 mg/dL) in a treat-to-target fashion according to the titration guideline. Dose adjustments were considered daily based on the pre-prandial and bedtime SMPG on the previous day. The dose adjustments were -1 or +1 if the pre-prandial or bedtime plasma glucose was <4.0 mmol/L or >6.0 mmol/L respectively. Basal insulin dose adjustments were allowed when needed. Metformin treatment continued without changing the frequency or dose.
Period: Overall Study
Arm/Group | Faster Aspart | NovoRapid
Started | 345 | 344
Exposed | 341 | 341
Completed | 301 | 305
Not Completed | 44 | 39
Not completed — Other, Subject wanted HbA1c to be > 7% | 1 | 0
Not completed — Other, weight gain, hypoglycaemic events | 1 | 0
Not completed — Other, Subject moved out of the country | 0 | 1
Not completed — Withdrawal by Subject | 15 | 15
Not completed — Lost to Follow-up | 5 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Adverse Event | 1 | 4
Not completed — Death | 1 | 1
Not completed — Withdrawal Criteria | 20 | 15

BASELINE CHARACTERISTICS:
Population: Full analysis set included all randomized subjects.
Groups:
- Faster Aspart: At randomization, all subjects started on 4 units of mealtime faster aspart (bolus insulin) in combination with once-daily sc injection of insulin glargine (basal insulin) and metformin (oral) in a basal-bolus regiment. Faster aspart was administered (sc) 0-2 minutes before each main meal and dose was titrated to the pre-prandial glycaemic target of 4.0-6.0 mmol/L (71-108 mg/dL) in a treat-to-target fashion according to the titration guideline. Dose adjustments were considered daily based on the pre-prandial and bedtime SMPG on the previous day. The dose adjustments were -1 or +1 if the pre-prandial or bedtime plasma glucose was <4.0 mmol/L or >6.0 mmol/L respectively. Basal insulin dose adjustments were allowed when needed. Metformin treatment continued without changing the frequency or dose.
- Total: Total of all reporting groups
Arm/Group | Faster Aspart | NovoRapid | Total
Number analyzed (Participants) | 345 | 344 | 689
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 241 | 248 | 489
  >=65 years | 104 | 96 | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (9.3) | 59.4 (9.6) | 59.5 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 171 | 353
  Male | 163 | 173 | 336
Glycosylated haemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin] | 7.96 (0.68) | 7.89 (0.71) | 7.92 (0.70)
Body Weight [Mean (Standard Deviation); unit: Kg] | 89.0 (16.9) | 88.3 (16.7) | 88.7 (16.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c
Description: The primary endpoint was change from baseline in HbA1c after 26 weeks of randomized treatment. For this endpoint baseline (week 0) and week 26 have been presented, where week 26 data is end of trial containing last available measurement.
Time Frame: Week 0, Week 26
Population: The analysis of this efficacy endpoint was based on the full analysis set (FAS). FAS included all randomized subjects. The statistical evaluation of the FAS was to follow the intention-to-treat (ITT) principle and subjects contributed to the evaluation 'as randomized'.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 345 | 344
Percentage of glycosylated haemoglobin
  Baseline (week 0) | 7.96 (0.68) | 7.89 (0.71)
  Week 26 | 6.63 (0.88) | 6.59 (0.84)
Statistical Analysis 1: Comparison: Faster Aspart vs NovoRapid; Change from baseline in HbA1c is analysed using a mixed-effect model for repeated measurements including changes from baseline in HbA1c at visit 14, 18, 22, 26, 30 and 36. The model includes treatment, region and continuous glucose monitoring (CGM) strata as fixed effects, subject as random effect, HbA1c at baseline as covariate and interaction between all fixed effects and visit, and between the covariate and visit; Test type: Non-Inferiority or Equivalence — The assessment was done by comparing the difference of faster aspart vs. NovoRapid®/NovoLog® in change from baseline in HbA1c after 26 weeks of randomized treatment to a non-inferiority limit of 0.4%; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.15 to 0.10] — The estimated parameter i.e mean difference is the estimated treatment difference for Faster aspart vs. NovoRapid (Faster aspart - NovoRapid)

2. Secondary Outcome: Change From Baseline in 2-hour PPG Increment (Meal Test)
Description: For this endpoint baseline (week 0) and week 26 have been presented, where week 26 data is end of trial containing last available measurement.
Time Frame: Week 0, week 26
Population: This endpoint was summarized using the Full Analysis Set (FAS). FAS included all randomized subjects.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 345 | 344
mmol/L
  Baseline (week 0): number analyzed (Participants) | 338 | 331
  Baseline (week 0) | 7.57 (3.19) | 7.34 (3.12)
  Week 26: number analyzed (Participants) | 342 | 342
  Week 26 | 4.55 (3.13) | 4.9 (3.36)

3. Secondary Outcome: Number of Treatment Emergent Confirmed Hypoglycaemic Episodes
Description: A hypoglycaemic episode was defined as treatment-emergent if the onset of the episode was on or after the first day of exposure to randomized treatment and no later than 1 day after the last day of randomized treatment. A severe or blood glucose (BG) confirmed hypoglycaemic episode was an episode that was severe according to the American Diabetes Association (ADA) classification (an episode that required assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a plasma glucose value <3.1 mmol/L (56 mg/dL) with or without symptoms consistent with hypoglycaemia.
Time Frame: From Week 0 to Week 26.
Population: This endpoint was summarized using the safety analysis set. Safety analysis set included all subjects receiving at least one dose of the test product or comparator. Subjects in the safety analysis set contributed to the evaluation 'as treated'.
Measure: Number; unit: Number of episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 341 | 341
Number of episodes | 2857 | 2692

4. Secondary Outcome: Change From Baseline in Body Weight
Description: as for outcome 2
Time Frame: Week 0, week 26
Population: This endpoint was summarized using the FAS. FAS included all randomized subjects.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 345 | 344
Kg
  Baseline (week 0) | 89.0 (16.9) | 88.3 (16.7)
  Week 26 | 91.6 (18.2) | 90.8 (17.7)

ADVERSE EVENTS:
Time Frame: All treatment-emergent adverse events (AEs) were collected from the date on or after the first day of exposure to randomized treatment until no later than 7 days after the last day of randomised treatment
Description: Safety analysis set was used for the assessment of safety including AEs. The safety analysis set included all subjects who received at least one dose of test product (faster aspart) or comparator(NovoRapid).
Arm/Group | Faster Aspart | NovoRapid
Serious Adverse Events (participants affected / at risk) | 15/341 | 24/341
Other Adverse Events (participants affected / at risk) | 49/341 | 53/341
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faster Aspart (N=341) | NovoRapid (N=341)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Arteriogram coronary (Investigations) | 0 (0) | 1 (1)
Aural polyp (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Carotid artery occlusion (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (4) | 3 (5)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Refractory anaemia with an excess of blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Wrong drug administered (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faster Aspart (N=341) | NovoRapid (N=341)
Nasopharyngitis (Infections and infestations) | 17 (20) | 24 (27)
Upper respiratory tract infection (Infections and infestations) | 16 (19) | 22 (27)
Urinary tract infection (Infections and infestations) | 20 (27) | 13 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more public disclosures may be prepared collaboratively by the Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.